CLINICAL TRIAL: NCT01748929
Title: Postpartum Deworming: Improving Breastfeeding and Optimizing Infant Growth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Theresa Gyorkos, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-198-GEN
Record Dates: First submitted 2012-12-07; First posted 2012-12-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Intestinal Diseases, Parasitic
Keywords: Global Health; Deworming; Postpartum; Soil-Transmitted Helminths; Pregnant Women
MeSH Terms: conditions — Intestinal Diseases, Parasitic | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albendazole (Experimental): single dose 400 mg tablet of albendazole
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): Placebo Manufactured by Hersil Laboratories in Lima, Peru
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole
  Arms: Albendazole
Drug: Placebo
  Arms: Placebo

SUMMARY:
Women of reproductive age are considered a high-risk group for worm infections by the World Health Organization. Maternal infection and anemia contribute to infant malnutrition by affecting milk quality and quantity, and duration of exclusive breastfeeding. To date, no study has investigated the health benefits of postpartum deworming to infants or mothers. A randomized controlled trial will be conducted in Peru to investigate the effectiveness of integrating deworming into routine postpartum care. The primary measure of effect will be infant weight gain between birth and six months of age. Other infant and maternal health indicators will also be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* Deliver at Hospital Iquitos
* Plan to reside in Iquitos or neighbouring area for the next 24 months
* Able to communicate in Spanish

Exclusion Criteria:

* Deliver multiples
* Delivery a stillborn or an infant with a serious congenital medical condition
* Transfered to another hospital prior to discharge

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Mean (± standard deviation) weight gain (kg) | Change between birth and six months of age

SECONDARY OUTCOMES:
Infant morbidity | 1, 6, 12, 24 months following birth
Maternal hemoglobin levels and anemia | 1, 6, 12, 24 months following birth
Breastfeeding practices | 1, 6, 12, 24 months following birth
  The prevalence of current, exclusive, predominant and partial breastfeeding will be used to assess breastfeeding practices. In accordance with WHO criteria, infants will be considered as exclusively breastfed if they ingest only breast milk (excluding vitamins and medications); considered as predominantly breastfed if, in addition to breast milk, they also ingest water, juice, teas, vitamins or medications, and considered as partially breastfed if their primary nutrition source is other than breast milk.
Maternal energy levels | 1, 6, 12, 24 months following birth
  Maternal energy levels will be measured using an adapted 5-item version of the Fatigue Assessment Scale (FAS) (Michielsen et al. 2004). This scale assesses symptoms of physical and cognitive fatigue.
Maternal STH infection | 1 and 6 months following birth
Breast milk quality | 1 and 6 months following birth
  Mean concentrations of key breast milk quality indicators (i.e. macronutrients, immunological factors, vitamins, and minerals) will be used to assess breast milk quality.
Breast milk quantity transferred from mother to infant | 1 and 6 months following birth

CONTACTS AND LOCATIONS:
Overall Officials: Theresa W Gyorkos, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Martin Casapia, MD, MPH, Principal Investigator — Asociación Civil Selva Amazónica
Locations (1):
- Asociación Civil Selva Amazónica, Iquitos, Peru

REFERENCES:
- [Derived] Mofid LS, Casapia M, Aguilar E, Silva H, Montresor A, Rahme E, Fraser WD, Marquis GS, Vercruysse J, Allen LH, Blouin B, Razuri H, Pezo L, Gyorkos TW. A Double-Blind Randomized Controlled Trial of Maternal Postpartum Deworming to Improve Infant Weight Gain in the Peruvian Amazon. PLoS Negl Trop Dis. 2017 Jan 5;11(1):e0005098. doi: 10.1371/journal.pntd.0005098. eCollection 2017 Jan. PMID 28056024
- [Derived] Mofid LS, Casapia M, Montresor A, Rahme E, Fraser WD, Marquis GS, Vercruysse J, Allen LH, Gyorkos TW. Maternal Deworming Research Study (MADRES) protocol: a double-blind, placebo-controlled randomised trial to determine the effectiveness of deworming in the immediate postpartum period. BMJ Open. 2015 Jun 17;5(6):e008560. doi: 10.1136/bmjopen-2015-008560. PMID 26084556